CLINICAL TRIAL: NCT03033017
Title: Predictors of Time to Viremia With an Analytic Treatment Interruption
Status: Withdrawn | Type: Observational
Why Stopped: Funding c hange
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 24777
Record Dates: First submitted 2016-10-07; First posted 2017-01-26 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lymph node biopsy: Inguinal lymph node biopsies will be collected per institutional guidelines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected on antiretroviral therapy 2 years: HIV-infected participants who have been on antiretroviral therapy (ART) for at least two years.
  Interventions: Other: Blood Testing

INTERVENTIONS:
Other: Blood Testing

SUMMARY:
This is a two-center study of 30 HIV-infected participants who have been on antiretroviral therapy (ART) for at least two years.

Participants will be asked to undergo LN and GALT biopsies both before and after a closely monitored analytic treatment interruption (ATI).

DETAILED DESCRIPTION:
The HIV field has made a dramatic shift to an emphasis on finding a cure for HIV.

However, there is no agreed upon test of cure, or even what the definition of a cure might be. The investigator believes the most reliable test of cure will be an analytic treatment interruption (ATI) with time to viremia as a standard measure of the impact of an intervention on the degree to which the reservoir has been depleted. This is rational as modeling studies utilizing ATI data point to reservoir size as an important predictor of time to viremia(1) and other studies have shown that levels of HIV DNA(2) and cell associated HIV RNA(3) prior to starting antiretroviral therapy (ART) are associated with time-to-rebound. However, these studies used a limited sampling strategy to determine when viremia rebounded and it is likely that greater sensitivity in measures of time-to rebound will be needed to accurately assess the impact of an intervention. The investigators have tested an ATI strategy where plasma HIV is sampled three times each week and ART is resumed once the virus becomes detectable. In this small, pilot study, the investigators sampled lymph nodes, GALT, plasma, and PBMC before, during, and after the ATI and found the time-to-rebound was 14 days (range 5 to 30 days) and that total years of ART exposure was associated with the time-to-rebound (4). The investigators propose a similar study that includes more intensive blood and lymphoid tissue sampling to identify factors that predict time to-rebound to provide a necessary foundation for future studies that utilize a treatment interruption as a test of efficacy for curative interventions.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected individuals who have been on ART therapy for at least two years
2. Male or Female, aged 18 years or older
3. Documented evidence of CD4+ T cell count ≥ 300 cells/µl for 12 months prior to study entry
4. BMI ≤ 30 or evidence by ultrasound or physical exam of peripheral inguinal lymph node(s) that is/are surgically accessible
5. Documented plasma HIV RNA levels below level of quantification <20 to <40 copies RNA/mL depending on the assay) ≥ 24 months (a single measurement above the level of detection but < 200 copies/ml will be allowed)
6. Willing to switch to an ART regimen consisting of dolutegravir and either tenofovir/emtricitabine or abacavir/lamivudine to avoid drugs with a long-half life that would expose the participant to a period of mono-therapy when the drugs are stopped.
7. Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during protocol
8. Able to provide voluntary written consent.

Exclusion Criteria

1. ART was initiated during acute infection (within first 6 months of infection)
2. Planning or current pregnancy or breastfeeding
3. History and/or presence of any clinically significant disease or disorder, such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disease/disorder, which, in the opinion of the enrolling physician, may put the participant at risk because of participation in the study, influence the results of the study, or affect the participant's ability to participate in the study.
4. Inability to comply with study procedures per enrolling physician discretion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 HIV-infected participants who have been on antiretroviral therapy (ART) for at least two years.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Time to viremia | Baseline to 14 days
  Time to viremia
Change in vRNA+ and vDNA+ cells | Baseline to 14 days
  measured by in situ hybridization and using quantitative image analysis to determine the frequency of + cell/gram lymphoid tissue
SCA (Single Copy Assay) | Baseline to 14 days
  performed as described in the protocol and reported as number of cells/ml plasma.
Change in markers of immune activation | Baseline to 14 days
  All measurements are the same IL1B, TNF, IL4, IL13, IL17, IL21,IL22, IL6, IL10
Change in CD4 | Baseline to 14 days
Change in CD4/CD8 ratio | Baseline to 14 days
Polyadenylation-RT-ddPCR assay for total transcripts (TAR) | Baseline to 14 days
  transcripts/million cells
ddPCR assays for read-through, elongated, polyadenylated, and multiply-spliced (Tat-Rev) transcripts | Baseline to 14 days
  reported as transcripts/million cells

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of California, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided